CLINICAL TRIAL: NCT03266484
Title: Effect of Dietary Therapy With a Probiotic Mixture on the Gut Microbiome and Fatigue Symptoms in Patients With Quiescent Inflammatory Bowel Disease - A Clinical Trial
Brief Title: Effect of a Probiotic Mixture on the Gut Microbiome and Fatigue in Patients With Quiescent Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Winclove Bio Industries BV (Industry)
Responsible Party: Principal Investigator, Ashwin Ananthakrishnan, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2017P001489
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: Microbiome; Fatigue; Probiotics
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Will be a double blinded randomized controlled trial. Masking will be done by the provider of the probiotics/placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic Mixture (Active Comparator): Participants who are meeting the inclusion criteria will be randomized to either the probiotic mixture or an identical placebo.
  The probiotics sachets will be taken twice a day for 12 weeks.
  Interventions: Dietary Supplement: Probiotic Mixture
- Placebo (Placebo Comparator): Participants who are meeting the inclusion criteria will be randomized to either the probiotic mixture or an identical placebo
  The identical placebo sachets will be taken twice a day for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Mixture — The probiotic supplement contains 8 different strains of bacteria and participants will be dosed in two dosages per a total of 40 billion bacteria daily.
  Arms: Probiotic Mixture
Dietary Supplement: Placebo — A placebo which is identical to the probiotic mixture. Participants will be dosed in two dosages daily.
  Arms: Placebo

SUMMARY:
The study is proposed as a single-site randomized double-blind placebo-controlled trial requiring 4 study visits, where two of the visits are combined with their appointment for routine clinical care. The study population will consist of patients with quiescent CD and UC and IBD-unspecified recruited from the Massachusetts General Hospital Crohn's and Colitis center. All eligible subjects will have a confirmed diagnosis of CD, UC, or IBD-unspecified according to accepted clinical, endoscopic, radiologic, and histologic criteria. Eligible patients will be contacted at the time of their routinely scheduled office visit and consented for the study. Self-report and review of medical records will be used to obtain detailed information regarding their disease on an intake questionnaire completed by a research study coordinator.

The study is proposed as a 12-week double-blind randomized controlled trial of the probiotic supplement compared to placebo. We propose to examine the effect of a specific probiotic supplement on the changes in the gut microbiome, serum metabolomic profile, and fatigue symptoms in patients with quiescent IBD.

Within 2 weeks of screening, eligible patients will be invited to visit MGH for a baseline visit. The patient will receive either the probiotic supplement or placebo for 4 weeks.

The first follow up visit will be at week 4 to check for adverse events on study treatment, to check accountability of probiotics/placebo, and to complete the set of questionnaires. Also, subjects will receive probiotic/placebo samples for the remaining 8 weeks of treatment.

At week 8, subjects will receive a phone call from a study research coordinator to check in with probiotics/placebo intake for treatment compliance and accountability records, and to complete the set of questionnaires ascertaining subjective symptoms.

Last study visit will be at week 12 which is often combined with a regular office appointment. Subject will provide serum blood and stool sample, as well as complete the set of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Confirmed CD or UC or IBD-unspecified diagnosed according to standard criteria
* Quiescent disease defined as Harvey Bradshaw index < 4 at baseline (week 0) or SCCAI < 2
* Persistent ongoing fatigue symptoms
* Endoscopic or radiologic remission within 12 months of screening
* Washout of non-study probiotic supplements for at least 4 weeks prior to screening.

Exclusion Criteria:

* Patients with clinical or endoscopically active inflammatory bowel disease
* Significant non-IBD comorbidity contributing to the fatigue (such as active cancer).
* Untreated severe depression or anxiety
* Known sleep disorders without adequate treatment,
* Presence of J-pouch or a stoma
* Ongoing use of other non-study probiotics
* Women who are pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change in gut microbiome | Week 12
  Change in fecal microbiome pattern assessed using 16sRNA sequencing.
Change in serum inflammatory cytokines levels | Week 12
  Change in inflammatory cytokines will be performed using the Biosciences Cytometric Bead Array kits.
Change in metabolomic profiles | Week 12
  Change in metabolic profiling will be performed on serum samples using established targeted quantitative and semi-quantitative gas chromatography-mass spectrometry (GC-MS) and liquid chromatography-mass spectrometry (LC-MS) methods
Change in fatigue symptoms | Week 4 and Week 12
  Reduction of fatigue symptoms which will be assessed using FACIT-F questionnaire. FACIT-F score of >43 at week 4 or week 12

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin N Ananthakrishnan, MBBS, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Crohn's and Colitis Center, MGH, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No